CLINICAL TRIAL: NCT06394466
Title: Evaluation of Thyroid Function and Autoimmunity in Subfertility Women and Thyroid Hormone Levels in the First Trimester of Assisted Reproduction
Brief Title: Thyroid Function and Autoimmunity in Subfertility Women and Assisted Reproductive Therapy
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Yuri Ian Lima Alves de Oliveira, M.D., Rio de Janeiro State University
Other Study IDs: Y201420y
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Failure; Thyroid Diseases
Keywords: Anti mullerian hormone; Thyroid autoimmunity; Antithyroid antibodies; Infertility
MeSH Terms: conditions — Thyroid Diseases; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing ovarian stimulation in our ART clinic: Inclusion criteria were: women attended in the outpatient clinic with baseline exams before ART and during ovarian stimulation between July 2021 and July 2023. Exclusion criteria were: patients with known clinical hypothyroidism, patients using medications that may influence the hypothalamic-pituitary-thyroid axis, such as glucocorticoids in supraphysiological doses; or that could interfere with thyroid hormone metabolism (lithium, amiodarone and aspirin in anti-inflammatory dosages).
  Interventions: Other: Non Applicable

INTERVENTIONS:
Other: Non Applicable — Non Applicable

SUMMARY:
The assessment of ovarian reserve is well established based on the dosage of anti-Mullerian hormone (AMH). The clinical applicability of detecting thyroid autoantibodies levels has been discussed as a potential marker of low-grade inflammation. There are no studies about the detection of these autoantibodies in infertile women. Our objective is to evaluate the association between ovarian reserve and thyroid function and its autoimmunity in infertile women seeking for assisted reproductive treatment (ART).Evaluation ot thyroid function in the first trimester in also be evaluated in women submitted to ART.

DETAILED DESCRIPTION:
The assessment of ovarian reserve is well established based on the dosage of anti-Mullerian hormone (AMH). The clinical applicability of detecting thyroid autoantibodies levels has been discussed as a potential marker of low-grade inflammation. There are no studies about the detection of these autoantibodies in infertile women. Evaluation of TSH profile during ovarian stimulation in ART is also debated in literature with conflicting results. Our objective is to evaluate the association between ovarian reserve and thyroid function and its autoimmunity in infertile women seeking for assisted reproductive treatment (ART) and TSH profile during ovarian stimulation and during the first trimester.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: women attended in the outpatient clinic with baseline exams before ART and during ovarian stimulation between July 2021 and July 2023

Exclusion Criteria:

* Exclusion criteria were: patients with known clinical hypothyroidism, patients using medications that may influence the hypothalamic-pituitary-thyroid axis, such as glucocorticoids in supraphysiological doses; or that could interfere with thyroid hormone metabolism (lithium, amiodarone and aspirin in anti-inflammatory dosages).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who looked for assisted reproduction and went through the process of ovarian stimulation and oocyte retrieval. The study was carried out with data from the first initial clinic appointment at Vida Assisted Reproduction clinic - Fertility Center (Rio de Janeiro, Brazil). Data collected from the patients in the initial clinical history were: chronological age, cause(s) of infertility, comorbidities and use of medications.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
TSH levels during assisted reproductive therapy and first trimester | 90 days
  TSH, free and total thyroxine, and ioduria in the first trimester

SECONDARY OUTCOMES:
Association between AMH levels and detectable categories of TPO-Ab or Tg-Ab | 30 days
  AMH, TPO-Ab and Tg-Ab dosages
Correlation between AMH and TSH | 30 days
  AMH and TSH dosages

CONTACTS AND LOCATIONS:
Overall Officials: Ana BW Tavares, pHD, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Vida Assisted Reproduction clinic - Fertility Center, Rio de Janeiro, Rio de Janeiro, Brazil